CLINICAL TRIAL: NCT02096822
Title: Efficacy of Facilited Tucking and Non-nutritive Sucking of Sterile Water to Relieve Preterm Infants From Pain During Heel-stick Procedures.
Brief Title: Efficacy of Facilitated Tucking During Pain Procedure in Preterm Infants
Acronym: BABYDOUL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: K13802; PHRI 13335 (Other: Assistance publique)
Record Dates: First submitted 2014-03-24; First posted 2014-03-26 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Facilitated Tucking; Non Nutritive Sucking; Preterm; Pain Relief
Keywords: Facilitated tucking; Non nutritive sucking; Preterm; Pain relief
MeSH Terms: conditions — Premature Birth | interventions — Facilitated Tucking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- non-nutritive sucking alone (Active Comparator): After randomization, baby will receive heel stick procedure with non-nutritive sucking and sterile water.
  Interventions: Other: non-nutritive sucking
- Facilitated tucking + non-nutritive sucking (Experimental): After randomization, baby will receive heel stick procedure with non-nutritive sucking and sterile water combined with facilited tucking.
  Interventions: Behavioral: Facilitated tucking + non-nutritive sucking

INTERVENTIONS:
Behavioral: Facilitated tucking + non-nutritive sucking
  Arms: Facilitated tucking + non-nutritive sucking
Other: non-nutritive sucking
  Arms: non-nutritive sucking alone

SUMMARY:
Preterm infants undergo very frequent painful procedures during neonatal care particularly during the first few days. The support for the pain of the preterm is a priority for nurses and neonatologists. Previous studies showed that non-nutritive sucking combined with sucrose ensures effective pain-relief for preterm (28-32 weeks GA). Unfortunately, the use of sucrose is limited to 4 administrations per day which is insufficient compared to the average of daily painful procedures. So, validation of an effective non-pharmacological intervention to relieve or avoid pain is essential. Facilitated tucking alone has been validated for preterm less than 37 GA during heel stick procedure with the PIPP score but no study looks for the benefit for pain relief of the association of non-nutritive sucking and facilitated tucking during heel stick procedure.

DETAILED DESCRIPTION:
After randomization, baby will receive heel stick procedure with either non-nutritive sucking and sterile water or non-nutritive sucking and sterile water combined with facilited tucking. The sequence will be filmed. Evaluation of PIPP and DAN will be done after viewing by 3 independent experts. Each child will receive only one procedure.

ELIGIBILITY:
Inclusion Criteria:

* Newborn from 28 weeks to 31 weeks +6 days GA.
* Age from 0 to 48 hours of life.
* Admission in intensive care unit or neonatal unit.
* Need for more than 4 heel stick procedures per 24 hours.
* One parents's consent

Exclusion Criteria:

* Hemodynamic instability with initropic drug need.
* Therapeutic Hypothermia in context of neonatal asphyxia.
* Curarized child.
* Neurologic anomaly of contact/tonus.
* Lidocaine application during the 4 hours before the procedure

Max Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2014-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
PIPP (Premature Infant Pain Profile) | 15 sec before to 30 sec after heel-lance procedure
  Behavioural measure of pain for premature infants.
  Indicators:
  * gestational age
  * behavioural state before painful stimulus
  * change in heart rate during painful stimulus
  * change in oxygen saturation during painful stimulus
  * brow bulge during painful stimulus
  * eye squeeze during painful stimulus
  * nasolabial furrow during painful stimulus

SECONDARY OUTCOMES:
DAN (Douleur Aigue Nouveau-né) | 15 sec before to 3 min after heel-lance procedure
  Behavioural measure of pain for premature infants
  Indicators:
  Facial movement Members movement Vocal expression

CONTACTS AND LOCATIONS:
Overall Officials: Anne Perroteau, Nurse, Principal Investigator — Assistance Publique
Locations (1):
- Hôpital A.Trousseau La roche Guyon, Paris, France